CLINICAL TRIAL: NCT07395167
Title: Evaluation of Soft Tissue Response and Prosthetic Complication of Three Different Provisional Prosthesis Used for Immediate Load Full Arch Implant Prosthesis. Randomized Control Clinical Trial
Brief Title: This Study Aims to Evaluate the Soft Tissue Response and Prosthetic Complications Associated With Three Different Types of Provisional Prosthesis Used in Immediate Loading Full-arch Implant Prosthetic Treatment. The Patients Are Randomly Assigned to the Three Groups to Compare the Clinical Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A08012024RP
Record Dates: First submitted 2026-01-10; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2023-12

CONDITIONS: Immediate Provisional Prosthesis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Printed provisional (Experimental): patients received 3D printed provisional full arch prosthesis
  Interventions: Device: 3D printed provisional full arch prosthesis
- Bar reinforced provisional (Experimental): patients received Bar reinforced 3D printed provisional full arch prosthesis.
  Interventions: Device: Bar reinforced 3D printed provisional full arch prosthesis
- Milled provisional (Experimental): patient received Milled PMMA provisional full arch prosthesis.
  Interventions: Device: Milled PMMA provisional full arch prosthesis

INTERVENTIONS:
Device: 3D printed provisional full arch prosthesis — patients received 3D printed provisional full arch prosthesis after implant placement
  Arms: Printed provisional
Device: Bar reinforced 3D printed provisional full arch prosthesis — patients received bar reinforced 3D printed provisional full arch prosthesis after implant placement
  Arms: Bar reinforced provisional
Device: Milled PMMA provisional full arch prosthesis — patients received Milled PMMA provisional full arch prosthesis after implant placement
  Arms: Milled provisional

SUMMARY:
This study aims to evaluate the soft tissue response and prosthetic complications associated with three different types of provisional prostheses used in immediate loading full-arch implant prosthetic treatment. The patients are randomly assigned to the three groups to compare the clinical outcomes and determine which provisional prosthesis provides better soft tissue health and fewer prosthetic complications

ELIGIBILITY:
Inclusion Criteria:

- In good general health. Controlled systemic diseases such as well-managed diabetes or hypertension. Good oral hygiene Adequate bone quality and quantity (Type I-III bone, ≥10mm height, ≥6mm width).

Exclusion Criteria:

* Uncontrolled systemic diseases Bone insufficiency Active infection or periodontal disease. Pregnancy. Heavy smokers (>10 cigarettes/day). History of previous implant failure in the same site. Immunocompromised patients (e.g., HIV, recent radiation therapy

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
clinical evaluation of dental implant (bone Level) | 3 months
  Evaluation included alveolar bone level around implant which is evaluated using periapical x-rays comparing T0 (at implant insertion) to T1 ( at one and half month) and T2 (at three months ) measuring amount of bone resorption around implant

SECONDARY OUTCOMES:
modified plaque index | 3 months
  the Modified Plaque Index (MPI) to assess peri-implant biofilm at four surfaces using scores from 0 (no plaque) to 3 (abundant plaque) using periodontal probe.
the Modified Gingival Index (MGI) | 3 months
  evaluate peri-implant soft tissue inflammation, scored from 0 (healthy mucosa) to 3 (severe inflammation)
peri-implant probing depth (PD) | 3 months
  measured with pressure-sensitive probes, where an increase over time indicates possible bone loss, with an ideal sulcus depth of less than 5 mm to allow effective oral hygiene

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura university faculty of dentistry, Al Mansurah, Egypt